CLINICAL TRIAL: NCT05401539
Title: The Effect of the Operating Room Tour Watched With a 3D Virtual Headset on Children's Fear and Anxiety of Preoperative- A Randomized Controlled Study
Brief Title: Effect of Virtual Tour of the Operating Theater on Fear and Anxiety of Preoperative Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Duygu Karaarslan, Principal Investigator, pediatric nursing research assistant, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MCBU-KARAARSLAN; 2020-083 (Other Grant/Funding Number: Scientific Research Projects Commission)
Record Dates: First submitted 2022-05-23; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Preoperative Anxiety
Keywords: Child,fear,anxiety,operating theater tour,virtual reality

STUDY DESIGN:
Intervention Model Description: This randomized controlled and experimental study will be conducted in the pediatric surgery clinic of a university hospital. Randomization of the children will achieve by checking the children at the beginning of each week and on the day of surgery according to the planned surgery lists. The VR tour provided with a 360° video is prepared to make the child be acquainted with the preoperative preparation process.The VR tour video feature actual nurses and physicians working in the surgery clinic and operating theatre. A professional VR company will performe filming in the hospital's operating theatre. The VR video is then will turn into an app for mobile devices. The children will assign into the VR-Documentary Film Group, VR- Operating Theater Tour Group and Control Group. A parallel trial design will use. Cardboard VR glasses, a non-pharmacological approach and a 3D imaging method, will use by the children to watch the movies.
Who Masked: Participant, Outcomes Assessor
Masking Description: In the process of assignment of children into groups, randomization is achieved in the computer by stratifying them in terms of sex and age variables (https://www.randomizer.org/).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: VR- Operating Theater Tour Group (Experimental): The 7-minute operating theatre tour, which describes the preparation process for the surgery, covers the following process: 6-12-year-old children's leaving their room, entering the operating theatre, and meeting the surgery team after they are taken to the operating theatre. The tour ends in the postoperative recovery unit. The actual operating theatre tour also will include information about how and when the child would wear the surgical gown, and how he or she would go to the operating theatre. In order to shoot the operating theatre tour scenes in the most appropriate way, all the procedures to be applied to the children to be operated will observe by the researcher in the pre-, intra- and post-operative periods. The scenario created for the scene shots will reviewe by experts in the field of filming and the final version will decide. The children who will have surgery will watch the real operating theatre tour with the cardboard VR headset.
  Interventions: Device: Cardboard VR
- Group 2: VR- Documentary Film Group (Experimental): The children in this group will watch the 5-minute musical documentary film featuring farm animals suitable for their age group with a cardboard VR headset. This group will form as a parallel group to determine whether the VR-Operating theatre Tour or the VR- Documentary Film is more effective.
  Interventions: Device: Cardboard VR

INTERVENTIONS:
Device: Cardboard VR — Google Cardboard is a discontinued virtual reality (VR) platform developed by Google. Named for its fold-out cardboard viewer into which a smartphone is inserted, the platform was intended as a low-cost system to encourage interest and development in VR applications. To use the platform, users run Cardboard-compatible mobile apps on their phone, place it into the back of the viewer, and view content through the lenses. The parts that make up a Cardboard viewer are a piece of cardboard cut into a precise shape, magnets or capacitive tape, a hook and loop fastener, a rubber band, and an optional near field communication tag. Smartphone is inserted in the back of the device and held in place by the selected fastening device. A Google Cardboard-compatible app splits the smartphone display image into two, one for each eye, while also applying barrel distortion to each image to counter pincushion distortion from the lenses.The result is a stereoscopic image with a wide field of view.

SUMMARY:
Experiences such as hospitalization, medical or surgical procedures are stressful, complex and threatening, especially for children and their families. Among the first crisis symptoms that children are faced with are illness, hospitalization and surgery anxiety. There is a direct relationship between the fear and anxiety experienced by children and their parents during the pre-operative processes. Therefore, ensuring not only the psychological but also physiological preparation of both the children and their parents before the surgery is of great importance. In the hospital, applying distraction methods appropriate for the age period of children and conveying procedural information to them simultaneously are difficult and challenging. In such situations, in clinical settings, virtual reality technology can be used at any time and place without requiring extra workforce to eliminate or reduce children's fear and anxiety. Virtual reality applications, as a distracting therapeutic method, are a fun, calming, safe, accessible, effective and acceptable intervention that can be used for the management of acute pain, fear and anxiety in pediatric patients. Such applications can affect children visually, aurally and contextually. Because they are different from common distraction methods used by children such as reading books, playing with toys, watching television or movies, playing a two-dimensional video game or game console. Virtual reality (VR) is used to distract children's attention to reduce fear and anxiety before surgery. A VR tour of the operating theater can provide a realistic experience for children. The aim in this study was to investigate the effect of an actual operating theater tour which is watched by children aged 6-12 years wearing a 3D virtual headset on their fear and anxiety.

DETAILED DESCRIPTION:
For school-age children aged 6-12, hospitalization and surgery mean a process full of worries causing anxiety and fear. In the preoperative period, children may feel threatened by being in an unfamiliar environment, seeing unfamiliar faces with masks, hearing the alarm sounds of devices, being exposed to medical procedures, and experiencing parental separation and parental anxiety. Preoperative anxiety is an important issue in pediatric patients because postoperative anxiety is related to preoperative anxiety and anxiety experienced at the beginning of anesthesia. The success of the surgery in children is related not only to the importance of the techniques and skills applied but also to the pre-operative preparation of children and meeting their and their parents' care needs. Therefore, preparing the child for the operation appropriately, being aware of the causes of anxiety and taking preventive measures in the preoperative period are very important for the physiological health of children and their parents. If the child is prepared for the operation in accordance with the procedures in the pre-operative period, it prevents the child from experiencing behavioral and physiological symptoms of anxiety. In children who are psychologically affected in the postoperative period, maladaptive behavioral changes such as anxiety, eating and sleep disorders, nightmares, enuresis, and tantrums are observed during the preoperative period. As observed in several studies, children whose anxiety levels are high in the preoperative period experience more complications during the postoperative recovery period. In addition, such anxiety experienced by children in the preoperative period causes them to stay in hospitals for a longer time (prolongs their hospitalization) in the postoperative period, which increases the burden and costs of health care significantly. In a study, it was observed that distracting 4-10-year old children's attention with tablets and phones in the pre-operative period decreased their stress and postoperative delirium, and anxiety experienced by their parents, and increased their cooperation with health personnel during the induction of anesthesia. Therefore, relieving preoperative anxiety not with pharmacological methods with side effects and potential risks but with non-pharmacological methods is of great importance.The use of non-pharmacological methods in children has been determined to be effective and safe. When which approach is to be applied to children is decided, the child's age, cognitive status, coping mechanisms, skills to keep up with digital age and use the technology should be taken into consideration because today's digital technology not only affects the whole world but also affects and changes the lives of children. Educational multimedia applications, web-based programs, visual and auditory technological tools are used to reduce children's preoperative anxiety and to create a more enjoyable experience by distracting their attention. With the latest developments in technology, lively, immersive and virtual reality systems have been included in the pre-operative preparation training of especially pediatric patients. Virtual reality technology enables children and their parents to be acquainted with the physical environment such as the operating theatre and recovery area in hospital environments they have not been in previously. A virtual reality tour, which is shown to children in the operating theatre before they undergo anesthesia, enables them to have a realistic, actual and inexpensive experience.Two mechanisms explaining the effect of virtual reality on anxiety are described as "exposure to the environment" and "distraction".Recent studies conducted on this issue show that virtual reality, an immersive technology, is an effective intervention to reduce preoperative anxiety in children. In randomized control studies conducted to determine children's preoperative anxiety levels, it was determined that the anxiety levels of children who used virtual reality technology were significantly lower than were those who of children did not use such technology. Preparing the child psychologically and eliminating his or her fear and anxiety in the pre-operative period will reduce the amount of anesthesia during the operation and that of analgesics after the operation, and will accelerate the child's recovery and early discharge. This will also reduce parents' anxiety. Therefore, the pediatric nurse should make the child be acquainted with the operation process by providing information to the child and the parent within the preoperative preparation programs, and teach them coping strategies by supporting them with emotional expressions.

The hypotheses of the present study are as follows:

H1: The operating theatre tour shown to children with a 3D virtual headset before the operation reduces their fear and anxiety.

H2: A documentary shown to children with a 3D virtual headset before the operation reduces their fear and anxiety.

ELIGIBILITY:
Inclusion Criteria:

Children are included in the study if they are aged between 6 and 12 years; have surgery for the first time; have outpatient surgery and only one operation at a time; could speak Turkish.

Exclusion Criteria:

Children will exclude in the study if they have genetic or congenital disease, have a chronic disease, and have previous surgery

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Information Form | in the preoperative period. it will take approximately 10-15 minutes to fill out the form.
  The Sociodemographic Information Form will administere to the children aged 6-12 years who will meet the inclusion criteria and their parents and agreed to participate in the study on the morning of the surgery day.

SECONDARY OUTCOMES:
Determining the preoperative anxiety scores of children | it will take approximately 10-15 minutes to fill out the form.
  in the preoperative period.
Determining the preoperative fear scores of children | it will take approximately 10-15 minutes to fill out the form.
  in the preoperative period.
Determining the preoperative anxiety scores of parents | it will take approximately 10-15 minutes to fill out the form.
  in the preoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical clinic of Manisa Celal Bayar University Hospital, Manisa, Turkey (Türkiye)